CLINICAL TRIAL: NCT01898715
Title: Phase 1 Study of the Safety and Tolerability of ATR-101 in Adrenocortical Carcinoma
Brief Title: Phase 1 Study of ATR-101 in Subjects With Advanced Adrenocortical Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millendo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATR-101-001
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Adrenocortical Carcinoma; Adrenal Cancer; ACC
Keywords: Adrenocortical carcinoma; Adrenal cancer; ACC
MeSH Terms: conditions — Adrenocortical Carcinoma; Adrenal Gland Neoplasms | interventions — N-(2,6-bis(1-methylethyl)phenyl)-N'-((1-(4-(dimethylamino)phenyl)cyclopentyl)methyl)urea hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATR-101 (Experimental): ATR-101 will be administered as capsules or tablets by mouth once or twice per day to ascending dose cohorts
  Interventions: Drug: ATR-101

INTERVENTIONS:
Drug: ATR-101

SUMMARY:
This first-in-human study is designed to establish the safety and tolerability of ATR-101 in patients with advanced adrenocortical carcinoma whose tumor has progressed on standard therapy. Information will also be collected to determine how long ATR-101 stays in the blood, and if any effect on tumor progression is seen. Biomarkers (blood and urine tests) will determine if any effects on production of steroid hormones (cortisol, aldosterone, estrogen and testosterone) are seen.

ELIGIBILITY:
Inclusion Criteria:

18 years;

* Clinical confirmation of adrenocortical carcinoma that is locally advanced or metastatic and not amendable to surgical resection;
* Failed or declined mitotane (adjuvant or therapeutic) therapy or a platinum-based chemotherapy regimen;
* Able to understand and comply with the protocol requirements;
* Willing and able to provide informed consent.

Exclusion Criteria:

* Mitotane level > 5
* Use of contraindicated concomitant medications
* Unstable medical condition that, in the judgment of the investigator, could interfere with study procedures or data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicity and determination of maximum tolerated dose | Occurrence of DLT at 28 days
  Adverse events will be recorded and tabulated by grade and system organ class according to CTCAE v 4.03. Laboratory measures and ECGs will be assessed.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of ATR-101 | Day 1 and Day 22
  Plasma levels of ATR-101 will be assessed after daily oral dosing and pharmacokinetic parameters will be calculated.
Change in plasma cortisol levels | Baseline and day 22
Change in objective measurement of tumor size | Baseline and 8 weeks
  CT or MRI scans will be read according to RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - National Institutes of Health/National Cancer Institute, Bethesda, Maryland
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - MDAnderson Cancer Center, Houston, Texas
- Comprehensive Cancer Center Mainfranken, University Hospital of Würzburg, Würzburg, Germany

REFERENCES:
- [Derived] Smith DC, Kroiss M, Kebebew E, Habra MA, Chugh R, Schneider BJ, Fassnacht M, Jafarinasabian P, Ijzerman MM, Lin VH, Mohideen P, Naing A. A phase 1 study of nevanimibe HCl, a novel adrenal-specific sterol O-acyltransferase 1 (SOAT1) inhibitor, in adrenocortical carcinoma. Invest New Drugs. 2020 Oct;38(5):1421-1429. doi: 10.1007/s10637-020-00899-1. Epub 2020 Jan 27. PMID 31984451
- [Derived] Lalli E, Sasano H. 5th International ACC Symposium: An Outlook to Current and Future Research on the Biology of Adrenocortical Carcinoma: Diagnostic and Therapeutic Applications. Horm Cancer. 2016 Feb;7(1):44-8. doi: 10.1007/s12672-015-0240-3. Epub 2015 Dec 14. PMID 26666256